CLINICAL TRIAL: NCT05616598
Title: Effect of New Oral Treatment for Hepatitis C Virus on Seminal Parameters
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Essam Mohamed El-sayed Akl, Assistant Professor of Dermatology and Andrology, Benha University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC 39-10-2022
Record Dates: First submitted 2022-11-01; First posted 2022-11-15 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Male Infertility; HCV
Keywords: Semen; DAA; Male infertility
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Intervention Model Description: DAA oral therapy for HCV.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pateint group (Active Comparator): Men with HCV
  Interventions: Drug: Sofosbuvir +daclatasvir+ simeprevir+Ribavirin
- Control group (No Intervention): Men without HCV

INTERVENTIONS:
Drug: Sofosbuvir +daclatasvir+ simeprevir+Ribavirin — Oral daily dose of Sofosbuvir +daclatasvir + simeprevir+ Ribavirin for 3 months
  Arms: Pateint group

SUMMARY:
Hepatitis C virus is commona viral infection. Direct-acting antiviral (DAA) oral drugs has been used in treatment of HCVs. the effect of these drugs on male infertility is still under investigation.

DETAILED DESCRIPTION:
Semen analysis will be done to male patients with HCV before and after treatment with DAA. The included men will take therapy for 3 months and HCV RNA titter will be evaluated. changes of seminal parameters will be recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

Men patients with HCV

Exclusion Criteria:

Patients with other hepatic disease, endocrinal disorder, malignancy, or urinary tract infection.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Men patients with HCV
Enrollment: 200 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Treatment of HCV | 3 months
  HCV titer by PCR is below detection level

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of Medicine, Benha University, Al Qalyūbīyah, Benha
  - Benha Faculty of Medecine, Banhā

IPD SHARING:
Plan to Share IPD: No